CLINICAL TRIAL: NCT06127524
Title: Biophysical Detection of Skin Changes to Cue Pressure Injury Prevention in Nursing Homes
Brief Title: Skin Change Actions by Nursing
Acronym: SCAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Duke University (Other); East Carolina University (Other); Boise State University (Other)
Responsible Party: Principal Investigator, Barbara Bates-Jensen, PhD, RN, FAAN, Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22-001256; 5R01NR020487-02 (NIH)
Record Dates: First submitted 2023-10-19; First posted 2023-11-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Pressure Injury
Keywords: Nursing homes; technology implementation; sub epidermal moisture
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: nursing home residents residing at any time in the facility during a 12 month baseline followed by 8 month intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Nursing Home Residents in intervention (Experimental): All Nursing Home residents in the facility during the 8 month intervention period
  Interventions: Device: SEM Scanner
- Nursing Home Residents in baseline (No Intervention): All Nursing Home residents in the facility during the 12 month baseline period

INTERVENTIONS:
Device: SEM Scanner — Implementation of the SEM Scanner as part of weekly standard skin assessments of sacrum and heels
  Other Names: Provizio SEM Scanner
  Arms: Nursing Home Residents in intervention

SUMMARY:
Pressure injuries, local areas of damage to the skin and underlying soft tissue that are costly and painful, are often preventable with timely use of prevention strategies. Identifying early pressure induced tissue damage among nursing home residents by nursing staff during routine skin assessment is critical for this process. Finding early damage can prompt nursing home staff to start prevention actions and may allow viable tissue rescue, reducing other health problems or death. We propose use of sub-epidermal moisture (SEM) measures as the cue for nursing home staff to start prevention care. SEM provides early detection of skin damage by as much as 5 to 10 days prior to other methods, eliminates the inherent structural bias in visual skin assessment for residents with dark skin tones, and demonstrates a model of care using technology innovation in poorly-resourced healthcare settings to provide bedside, real-time, point-of-care feedback that is can be used immediately by nursing staff.

In this study, nursing staff will use a device (the Provizio SEM Scanner) as part of standard skin assessments. The staff will use the values from the Provizio SEM Scanner during these assessments to decide if residents need preventive care for their skin. The study will look at these decisions and residents' subsequent health outcomes.

The study will also use information about residents' skin health and prevention actions during the 52 weeks before the study as a comparison.

DETAILED DESCRIPTION:
Pressure injuries (PrIs), commonly located over bony prominences, are local areas of damage to the skin and underlying soft tissue (often not initially visible) caused by pressure and shear forces. These costly injuries, up to $151,000 per PrI, are associated among nursing home (NH) residents with reduced quality of life, pain, depression, and mortality. Prevalence and incidence of PrI have not declined and facility-acquired PrIs (FAPrIs) have actually increased over the last decade in NHs despite use of standardized prevention care. In fact, nursing home FAPrI rates are nearly double (5.4%) hospital FAPrI rates (2.9%).For nursing staff, the standard method of detecting changes in skin is conducting a visual assessment for skin discoloration; this visual detection coupled with risk assessment, serve as the customary trigger for initiating PrI prevention strategies. However, by the time reddened skin (erythema) is detected, significant damage is already present. The lag time between skin change associated with PrI formation and visual detection of the change eliminates the potential for PrI prevention strategies to be effective. Furthermore, visualization of potential PrIs is complicated by the challenge of discerning discoloration on persons with dark skin tones which, makes NH residents from minority or under-represented racial/ethnic groups more at-risk, thus leading to a significant health disparity. Multiple studies have shown racial/ethnic health disparities in PrI prevalence and incidence, severity, time to development and healing In fact, disparities in PrI prevalence, when comparing Black and white NH residents, are pervasive and persistent. Early detection of skin and tissue changes occurring as a PrI develops is a fundamental component in effective implementation of PrI prevention protocols.

Technological advances in biophysical measures have strengthened the capacity to detect early changes in tissue characteristics, for any skin tone, thus facilitating prevention care. A subclinical PrI can be readily identified at the dermal, and muscle tissue layers with a biophysical approach. Measurement of subepidermal moisture (SEM) using surface electrical capacitance is one biophysical method that has been shown to detect and predict early pressure damage. The SEM Scanner, a device used to date only in acute care hospitals, provides a biophysical measure of local inflammation and edema related to early pressure damage with a numerical result that serves as a cue for nursing staff to initiate PrI prevention with subsequent successful reduction and sustained decline in FAPrI incidence occurring. This technology's effectiveness has been demonstrated in hospitals; and this study will be the first to extend the use to NHs, a setting that is low in resources and desperate for assistance in this area. An embedded pragmatic stepped wedge clinical trial design will be conducted in 6 NHs within a single NH company with standardized operating procedures and PrI prevention protocols. We will examine whether SEM assessment results reflecting detection of early pressure damage can serve as an effective cue for NH nursing staff initiation of PrI prevention actions with the goal of reducing FAPrI rates over a 8-month intervention period. Specific aims are to:

Aim 1. Determine if early pressure damage detected by SEM assessment at time of visual skin observation of NH resident sacral and heel areas is effective in cueing the initiation of NH standard PrI prevention.

Aim 2. Examine the association between NH standard PrI prevention and SEM assessment and NH residents' characteristics (age, gender, risk, skin tone, race, ethnicity, BMI, Cognitive status) and their interactions on individual NH residents with regard to initiation of PrI prevention and PrI occurrence.

Aim 3. Explore if SEM usability, NH, and nursing staff characteristics influence the adoption and assimilation of early PrI detection and subsequent PrI prevention practices.

Results from this study will increase our knowledge and advance PrI prevention science and nursing practice. Furthermore, the clinical utility and relevance achieved with real world testing and staff delivery will help NHs with high PrI incidence by adding to the clarity of preventive nursing practices. These results will also be used for developing specialty policies and guidelines like the international PrI prevention clinical practice guidelines.

ELIGIBILITY:
Nursing home residents:

Inclusion Criteria:

For intervention, must reside in nursing home at least 1 day during 8-month study period and be at least 18 years old at study start.

For baseline period: Must reside in nursing home at least 1 day during 52-week lookback period and be at least 18 years old at study start

Exclusion Criteria:

For intervention: Did not reside in nursing home during 8-month study period or younger than 18 years old For baseline period: Did not reside in nursing home during 52-week lookback period or younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4733 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
New pressure injury prevention initiated | From date of identified skin damage through 3 days later, assessed up to 8 months for intervention period or up to 12 months for baseline period
  At least one Pressure Injury Prevention action newly initiated defined as electronic health record (EHR) documentation

SECONDARY OUTCOMES:
Time to pressure injury prevention initiation | Number of days from date of identified skin damage through 3 days later, assessed up to 8 months for intervention period or up to 12 months for baseline period
  Number of Days from skin assessment until EHR documentation of Pressure Injury Prevention

OTHER OUTCOMES:
Sacral and/or heel pressure injury occurrence | From at least 3 weeks since prior pressure injury occurrence (if ever), assessed up to 8 months for intervention period or up to 12 months for baseline period
  EHR documentation of sacral and/or heel PrI
Time to pressure injury occurrence | Number of days from date of new pressure injury occurrence (from at least 3 weeks since prior pressure injury, if ever), assessed up to 8 months for intervention period or up to 12 months for baseline period
  Number of pressure injury free days since prior pressure injury occurrence, if ever.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M Bates-Jensen, PhD, Principal Investigator — Univeristy of California Los Angeles; Tracey L Yap, PhD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Large proprietary nursing home chain faciity #3, Kennett Square, Pennsylvania
  - Large proprietary nursing home chain facility #1, Kennett Square, Pennsylvania
  - Large proprietary nursing home chain facility #4, Kennett Square, Pennsylvania
  - Large proprietary nursing home chain facility #5, Kennett Square, Pennsylvania
  - Large proprietary nursing home chain facility #6, Kennett Square, Pennsylvania
  - Large proprietary nursing home chain facility #7, Kennett Square, Pennsylvania
  - Large proprietary nursing home chain facilty #2, Kennett Square, Pennsylvania

IPD SHARING:
Plan to Share IPD: No